CLINICAL TRIAL: NCT00315250
Title: Development of Imaging, Clinical and Biochemical Bio-Markers for Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Molecular NeuroImaging (Other)
Responsible Party: Principal Investigator, Danna Jennings, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Query 3C
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson's Disease; Parkinsonian Syndrome
Keywords: Parkinson
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [123I]β-CIT (Experimental): To assess B-CIT and SPECT imaging
  Interventions: Drug: [123I]β-CIT

INTERVENTIONS:
Drug: [123I]β-CIT — Single Photon Emission Computed Tomography
  SPECT imaging uses the single photon emissions from radioactive compounds that are (most commonly) injected into a patient and are metabolized by specific organs or body systems. SPECT imaging is performed by using a gamma camera to acquire multiple 2-D images (also called projections), from multiple angles. A computer is then used to apply a tomographic reconstruction algorithm to the multiple projections, yielding a 3-D dataset. This dataset may then be manipulated to show thin slices along any chosen axis of the body, similar to those obtained from other tomographic techniques, such as MRI, CT, and PET. The resulting SPECT images reflect body/organ function as opposed to specific anatomy of other imaging modalities such as CT or MRI.
  Other Names: SPECT imaging

SUMMARY:
We propose to build on preliminary data evaluating non-dopaminergic/non-motor clinical biomarkers to more fully assess these markers at the threshold of Parkinson disease (PD).

Development of reliable biomarkers for both dopaminergic and non-dopaminergic manifestations of Parkinson disease (PD) and related disorders may dramatically accelerate research on PD etiology, pathophysiology, and therapeutics. Biomarkers are broadly defined as characteristics that are objectively measured and evaluated as indicators of normal biological processes, pathogenic processes, or pharmacologic responses to a therapeutic intervention. Specific biomarkers may be useful at the onset of neurodegeneration, the onset of disease, and/or to mark disease progression.

DETAILED DESCRIPTION:
Two hundred patients who have undergone neurological evaluation by their general community neurologist and have a questionable diagnosis of PD will be recruited to participate in this study. Subjects will be referred by the neurologists to the Institute for Neurodegenerative Disorders (IND) in New Haven, CT.

All subjects will be clinically evaluated at IND by a two movement disorders experts. At the baseline visit all subjects will also undergo [123I]ß-CIT SPECT ANAM, voice acoustics, olfactory, Spiral and biochemical testing. Each movement disorders expert will make an initial clinical diagnosis at baseline and again within three months follow-up. At the three month visit one movement disorder expert will be provided the DAT imaging data and will review that data with the subjects and referral physician. The other movement disorders physician will remain blind to the imaging and all other biomarker data. The blinded movement disorders expert will provide a final clinical diagnosis at the 12 month follow-up visit, which will represent the 'gold standard' diagnosis in this study. Statistical analysis to determine the sensitivity and specificity of ANAM, voice acoustics, olfactory, Spiral and biochemical testing compared to [123I]ß-CIT SPECT, and the gold standard clinical diagnosis will be completed. All subjects with DAT deficit and 10% of those without DAT deficit will be asked to return for repeat evaluation at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Older than 21
* Any parkinsonian symptoms
* Referral by community neurologist
* Parkinsonian symptoms for less than 2 years duration.
* Willingness to follow the study plan.

Exclusion Criteria:

* Pregnancy
* Significant medical disease including abnormalities on screening biochemical or hematological labs or abnormal electrocardiogram (ECG - tracing of the electrical activity of the heart)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2006-01; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Assess the sensitivity and specificity of olfaction, upper limb kinematic behavior, cognition, voice, metabolomic, proteomic and gene expression profiling in categorizing Parkinson Syndrome (PS) vs non-PS | 2 years
  Assess the sensitivity and specificity of olfaction, upper limb kinematic behavior, cognition, voice, metabolomic, proteomic and gene expression profiling in categorizing Parkinson Syndrome (PS) vs non-PS defined by >30% age expected loss of [123I]B-CIT SPECT uptake.

SECONDARY OUTCOMES:
Assess sensitivity and specificity of olfaction, upper limb kinematic behavior, cognition, voice, metabolomic, proteomic and gene expression profiling in categorizing PS vs non-PS | 2 years
  Assess sensitivity and specificity of olfaction, upper limb kinematic behavior, cognition, voice, metabolomic, proteomic and gene expression profiling in categorizing PS vs non-PSby clinical exam by a movement disorders expert (blinded to any imaging data) after 12 months of subject follow up.
Correlate progression of biomarker outcomes for olfaction, upper limb kinematic behavior, cognition, voice, metabolomic and gene expression profiling with progression of PS defined by % change from baseline in putamen [123I]ß-CIT SPECT uptake. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States